CLINICAL TRIAL: NCT06980597
Title: An Open-Label, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Allogeneic CAR-T Cell Therapy (OL-108) in the Treatment of Relapsed/Refractory Autoimmune Diseases
Brief Title: A Study of OL-108 in Relapsed/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Kai Hu, Professor, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OL-108-001
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus (SLE); Idiopathic Inflammatory Myopathy (IIM); Systemic Sclerosis (SSc); ANCA Associated Vasculitis (AAV)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Myositis; Scleroderma, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OL-108 (Experimental)
  Interventions: Biological: OL-108

INTERVENTIONS:
Biological: OL-108 — OL-108 will be given through IV bolus with ascending dose levels to determine the maximum tolerated dose (MTD)

SUMMARY:
This study aims to characterize the safety, tolerability, pharmacokinetics, and preliminary efficacy of OL-108 in relapsed/refractory autoimmune diseases.

DETAILED DESCRIPTION:
This is an open-label, single-arm, clinical study to evaluate the efficacy and safety of CAR-T therapy OL-108 in the treatment of Relapsed/ Refractory Autoimmune Disease such as SLE, IIM, SSc and AAV.

ELIGIBILITY:
Inclusion Criteria:

* General:
* Adults aged 18-65 years old
* ECOG 0-2
* Adequate organ function
* Females of childbearing potential (FCBP) must have a negative pregnancy test at screening and must agree to use a highly effective contraceptive method starting from the time of lymphodepletion and for 2 years after dosing of the IMP
* SLE specific:

  a) Fulfilling the 1997 ACE SLE criteria/ 2012 SLICC criteria/ 2019 ACR/EULAR classification criteria of SLE; b) A positive ANA titer (≥ 1:80) and/or presence of anti-dsDNA, or anti-Sm antibodies; c) Active disease at screening, defined as SLEDAI-2K≥8 AND clinical SLEDAI-2K≥6, AND ≥1 organ system with a British Isles Lupus Assessment (BILAG) A score (severe disease activity) or ≥2 organ systems with a BILAG B score (moderate disease activity), AND PGA≥ 1; OR biopsy proven 2003 ISN/RPS class III/IV +/- class V lupus nephritis; d) relapsed or refractory to at least one immunosuppressant or biologic.
* IIM specific:

  a) Fulfilling the 2017 ACR/EULAR classification criteria for DM, PM, ADM, ASS and IMNM; b) Active disease as defined by at least one of the following criteria: at least one muscle enzyme > ULN in the past 4 weeks, active disease by EMG/muscle biopsy/MRI in the past 3 months, active DM rash; c)MMT < 142 and 2 of the following criteria: VAS patients Global ≥ 2 cm, VAS physician Global ≥ 2 cm, HAQ > 0.25, at least one muscle enzyme > 1.5x ULN, MDAAT ≥ 2 ; d) CDASI ≥14 if with skin involvement; e) At least one myositis-specific or associated antibody positive; f)relapsed or refractory to at least one immunosuppressant or biologic.
* SSc specific:

  a)Fulfilling the 2013 ACR/EULAR classification criteria of SSc; b) Active disease as defined by one of following: new or progressing skin manifestation/vital organ involvement within 6 months prior to screening, CRP≥6 mg/L, ESR≥28 mm/h, platelet ≥330 × 10⁹/L; c) mRSS score >10; d)relapsed or refractory to at least one immunosuppressant or biologic.
* AAV specific:

  1. Fulfilling the 2022 ACR/EULAR classification criteria for MPA/GPA; b) Presence of ANCA to either proteinase 3 or myeloperoxidase; c)At least one major or three non-major items or at least two renal items of hematuria and proteinuria on the BVAS; d)relapsed or refractory to at least one immunosuppressant or biologic.

Exclusion Criteria:

* Active uncontrolled infection
* Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy or with detectable HBV viral load
* Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load
* HIV antibody positive
* Syphilis antibody positive
* Active tuberculosis, untreated or inadequately treated latent tuberculosis infection (LTBI)
* History of serious infection within 3 months prior to screening (defined as requiring hospitalization or intravenous antimicrobial therapy), or history of oral antimicrobial therapy within 1 month prior to screening (e.g., viral infections, opportunistic infections, including but not limited to severe cytomegalovirus or herpes virus infections)
* Congenital long QT syndrome or a corrected QTcF interval of ≥480 ms at screening (unless secondary to pacemaker or bundle branch block)
* Uncontrolled hypertension (blood pressure ≥160/100 mm Hg repeatedly), unstable angina, congestive heart failure (greater than New York Heart Association class II), electrocardiographic evidence of acute ischemia, coronary angioplasty or myocardial infarction within 6 months prior to screening, uncontrolled atrial or ventricular cardiac arrhythmia, poorly controlled diabetes or other endocrine diseases, severe chronic pulmonary disease, or other serious medical condition which is likely to significantly impair the patient's ability to tolerate the study treatment
* history of organ transplant
* Pregnancy or lactating women
* Use of any other experimental medication within 4 weeks or 5 half-lives prior to start of study drug
* Use of biologics within 3 months, stem cell transplant or CAR-T within 6 months prior to the start of study drug
* Received live or attenuated vaccine within 4 weeks of Cycle 1 Day 1
* Presence of other autoimmune or auto-inflammatory diseases that may affect study assessments, such as rheumatoid arthritis, gout, or active fibromyalgia syndrome.
* Limited to patients diagnosed with SLE: patients with active neuropsychatric SLE
* Limited to patients diagnosed with IIM: Severe involvement of respiratory muscles affecting ventilatory function; permanent muscle weakness related to IIM; other inflammatory or non-inflammatory myopathy: inclusion body myositis, infectious myopathy, metabolic myopathy, muscular dystrophy or a family history of muscular dystrophy, drug-induced or endocrine-induced myositis, and juvenile myositis
* Limited to patients diagnosed with SSc: at risk for scleroderma renal crisis; SSc-associated gastric antral vascular ectasia; Severe gastrointestinal involvement leading to malabsorption or intestinal failure
* Limited to patients diagnosed with AAV: Central nervous system vasculitis; Alveolar hemorrhage requiring invasive pulmonary ventilation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | After OL-108 administration up to 30 days (Day 1-Day 30)
  Adverse events will be assessed based on the CTCAE 5.0
Treatment emergent adverse event (TEAE) incidence and severity | From lymphodepletion through study completion, up to 2 years
  Adverse events will be assessed based on the CTCAE 5.0

SECONDARY OUTCOMES:
Overall Response Rate | Baseline through study completion, up to 2 years
  The efficacy outcome variable, Overall Response Rate (ORR), is defined as the ratio between the number of subjects experiencing a response at weeks 12, 24 and 52 and the total number of enrolled subjects.
  A response to treatment will be considered as:
  * SLE: Fulfillment of DORIS remission/LLDAS criteria of SLE.
  * SSc: Fulfillment of mCRISS criteria
  * IIM: 2016 ACR/EULAR Total Improvement Score.
  * AAV: Birmingham vasculitis activity score (BVAS) of 0.
Cmax of OL-108 | Baseline through study completion, up to 2 years
  The maximum concentration of the CAR-T cells will be measured to assess OL-108 in vivo expansion and persistence.
Tmax of OL-108 | Baseline through study completion, up to 2 years
  The time of the maximum concentration will be measured to assess OL-108 in vivo expansion and persistence.
AUC 0-28 days of OL-108 | Baseline through study completion, up to 2 years
  Area under the curve will be measured to assess OL-108 in vivo expansion and persistence.
Serum cytokines | From lymphodepletion till day 90
  The levels of cytokines will be measured, such as IL-6 and ferritin.
Level of Immunogenicity | Baseline through study completion, up to 2 years
  To assess the presence of antibodies to OL-108 (ADA)
Level of RCR | Baseline through study completion, up to 2 years
  To determine whether Replication Competent Retrovirus (RCR) is present in patients that receive OL-108

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Boren Hospital, Beijing
  - Beijing GoBroad Hospital, Beijing